CLINICAL TRIAL: NCT05452174
Title: Endeavor to Stop Nausea/Vomiting Associated With Pregnancy (E-SNAP)
Acronym: ESNAP
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: transfer of PI to new organization
Sponsor: Northwestern University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00215676; R21HD105101 (NIH)
Record Dates: First submitted 2022-06-29; First posted 2022-07-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy; Severe Nausea and Vomiting; Hyperemesis Gravidarum
Keywords: pregnancy; severe nausea; vomiting
MeSH Terms: conditions — Nausea; Vomiting; Hyperemesis Gravidarum | interventions — Mirtazapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mirtazapine Treatment Arm (Experimental): Subjects will be administered the initial dose of mirtazapine, with dosage progressively increased over the course of the study. The initial dose of mirtazapine is 15 mg tablet, once per day. The dose will be increased weekly as tolerated up to 45 mg per day. The dose will be increased by 15 mg each week if the lower dose is tolerated without significant side effects. That is to say, the subject will take 15 mg/day every day for the first week, 30 mg/day every day for the second week, and 45 mg/day every day for the third week, with the option of the subject continuing the medication for the remainder of the pregnancy. If subjects choose to discontinue the mirtazapine, there will be a tapering regimen: if a patient is taking 45 mg at the end of week 3, they will begin a taper (by week) of 30 to 15 to 7.5 to 0 mg. If they relapse or has discontinuation symptoms, the previous effective dose will be given. They may attempt to taper again with the same approach.
  Interventions: Drug: Mirtazapine

INTERVENTIONS:
Drug: Mirtazapine — Mirtazapine, sold under the brand name Remeron, is an atypical antidepressant, and as such is used primarily to treat depression.
  Other Names: Remeron

SUMMARY:
The primary objective of this proposal is to conduct an early Phase 2 clinical trial to determine the acceptability, dosing, tolerability and safety of mirtazapine for severe nausea and vomiting of pregnancy (sNVP) that is not adequately responsive to current standard treatments. This plan mirrors clinical practice since commonly prescribed antiemetic/ antinauseant drugs will be tested for efficacy before treating with mirtazapine.

DETAILED DESCRIPTION:
Translational Research in Maternal and Pediatric Pharmacology and Therapeutics (PAR-20-299) supports research to "enhance the usage of existing drugs or drug repurposing for safer and more effective treatment for pregnant women" for "the early and conceptual stages of these projects. The primary objective of this proposal is to conduct an early Phase 2 clinical trial to determine the acceptability, dosing, tolerability and safety of mirtazapine for severe nausea and vomiting of pregnancy (sNVP) that is not adequately responsive to current standard treatments. This plan mirrors clinical practice since commonly prescribed antiemetic/ antinauseant drugs will be tested for efficacy before treating with mirtazapine.

Mirtazapine is a promising drug to repurpose for sNVP. It has potent anti-emetic properties and is available as an oral disintegrating formulation. It is used off-label to treat NV during cancer chemotherapy, prevent post-surgical nausea and vomiting and for gastroparesis. It is marketed as the serotonin-norepinephrine reuptake inhibitor antidepressant Remeron®. Mirtazapine has multiple receptor effects beyond those involved in reducing depressive symptoms. In cancer and chemotherapy patients, it produces rapid resolution of nausea and vomiting by blocking physiologic inputs that coordinate emesis. It is hypothesized that repurposing mirtazapine for obstetric use overcomes the challenges of traditional pathways to develop new agents because its pharmacokinetics, safety and dosing have been established for general populations of patients and exposure data are available because it is prescribed to pregnant persons with depression.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* inpatient or outpatient status
* English speaking
* obstetrician's evaluation and diagnosis of sNVP or HG
* tolerance of oral disintegrating tablet at bedtime
* PUQE score of 10-15; moderate/high or severe
* refractory sNVP
* blood pressure range 70-200 / 45-120
* normal ECG

Exclusion Criteria:

* allergic or adverse reaction to mirtazapine
* patient has bipolar disorder
* subjects with active depression, or history of or current active suicidal ideation or attempt
* subjects with renal or hepatic impairment
* substance about in last 6 months
* use of medicinal or recreational cannabis-derived products in the last 6 months
* taking MAOIs, strong CYP3A inducers or inhibitors, and SSRIs

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-10-29 (Actual); Study Completion 2023-10-29 (Actual)

PRIMARY OUTCOMES:
change in Pregnancy Unique Quality of Emesis (PUQE) score | daily for three weeks
  We will utilize the PUQE scale to capture the severity of nausea and vomiting in pregnancy based on three physical symptoms: nausea, vomiting, and retching over the previous 24 hours. A PUQE score of < 6 is considered mild, a score from 7-12 is moderate, and a score of 13+ is considered severe. This scale will be entered daily in REDCap directly by the participant.

SECONDARY OUTCOMES:
Self-Administered Comorbidity Questionnaire (SCQ) | weekly for three weeks
  The Comorbidity Questionnaire (CQ) assesses comorbid conditions in clinical and health services research. The questionnaire is self-administered, short, easily understood, and can be completed by individuals without any medical background. It also allows the subject to note the severity of each comorbid conditions and their perception of its impact on their function.
9-Item Patient Health Questionnaire (PHQ-9) | weekly for three weeks
  The 9-Item Patient Health Questionnaire (PHQ-9) is a self-administered instrument based on the nine DSM-5 criteria listed under criterion A for Major Depressive Disorder. The questionnaire includes criteria based diagnosis of depressive symptoms, assists in identifying treatment goals, determining severity of symptoms, as well as guiding clinical intervention. When considering a diagnosis, the clinician will use clinical interviewing skills to determine whether the symptoms are causing clinically significant distress or impairment and those symptoms are not better explained or attributed to other conditions, such as substance use, medical conditions, or bereavement.
Generalized Anxiety Disorder Scale, 7-item (GAD-7) | weekly for three weeks
  The Generalized Anxiety Scale is a 7-item self-report for symptoms consistent with the Diagnostic and Statistical Manual of Mental Disorders of generalized anxiety disorder.
Peripartum Events Scale (PES) | weekly for three weeks
  The Peripartum Events Scale (PES) captures data from several categories in the birth record. The following categories of events are included: medical and obstetric risk factors, time in operating room, fetal monitoring, surgical complications, infant anthropometrics and outcome, NICU admission, and postpartum complications (such as infection, hemorrhage). Admission to the special care nursery will also be noted. We have modified the original measure to align with current obstetrical practices. The PES will be completed for all enrolled participants.
PROMIS Global Health | weekly for three weeks
  The PROMIS Global Health item scale assesses overall health. The global health items include ratings of the five primary PROMIS domains (physical function, fatigue, pain, emotional distress, social health) as well as perceptions of general health that cut across domains.
Columbia-Suicide Severity Rating Scale (C-SSRS) | weekly for three weeks
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a questionnaire used for suicide assessment that was developed with NIMH support. The scale is evidence-supported and is part of a national and international public health initiative involving the assessment of suicidality. Suicidal ideation will be assessed at baseline, during, and 28 days after treatment cessation if there were any abnormalities during the trial.
plasma mirtazapine concentrations | weekly for three weeks
  Genotypes that determine the activities of CYP2D6, and minor pathways 3A4/5 and 1A2, will be explored for associations with mirtazapine plasma concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Wisner, M.D., M.S., Principal Investigator — Northwestern University (adjunct) now at Children's National Hospital
Locations (1):
- Northwestern University Asher Center for the Study and Treatment of Depressive Disorders, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abramowitz A, Miller ES, Wisner KL. Treatment options for hyperemesis gravidarum. Arch Womens Ment Health. 2017 Jun;20(3):363-372. doi: 10.1007/s00737-016-0707-4. Epub 2017 Jan 9. PMID 28070660
- [Background] Fejzo MS, MacGibbon KW, Wisner KL. Pregnant, miserable, and starving in 21st century America. AJOG Glob Rep. 2022 Dec 5;3(1):100141. doi: 10.1016/j.xagr.2022.100141. eCollection 2023 Feb. PMID 36536797

DOCUMENTS (3):
  • Study Protocol (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT05452174/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT05452174/SAP_001.pdf
  • Informed Consent Form (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT05452174/ICF_002.pdf